CLINICAL TRIAL: NCT06987708
Title: Evaluating the Impact of a 12-month Multi-Modal Lifestyle Management Intervention on Disease Relevant Biomarkers Associated With Monoclonal Gammopathy of Unknown Significance (MGUS) and Smoldering Myeloma (SM): A Prospective Intervention Pilot Study
Brief Title: Evaluating the Impact of a 12-month Multi-Modal Lifestyle Management Intervention on Disease Relevant Biomarkers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Center for Cancer Lifestyle Management (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MGUS-SM-Lifestyle; Pro2024-0235 (Other: HMH)
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Monoclonal Gammopathy of Uncertain Significance; Smoldering Myeloma
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multimodal Lifestyle Intervention (Experimental)
  Interventions: Other: The Multimodal Lifestyle Intervention

INTERVENTIONS:
Other: The Multimodal Lifestyle Intervention — The multimodal lifestyle intervention has six foci: positive cognition, exercise/movement, stress reduction, social connection, emotional well-being, and nutrition

SUMMARY:
A prospective, pilot study to assess the impact of a 12-month multi-focal lifestyle intervention on myeloma-relevant biomarkers in patients with MGUS or SM. The multimodal lifestyle intervention has six foci that patients will participate in over the course of one-year.

DETAILED DESCRIPTION:
Patients with a diagnosis of MGUS or SM who are willing and able to participate in this 12-month multimodal lifestyle approach. Eligible patients include those 18 years of age and older diagnosed with MGUS/SM, ECOG PS 0-2, absence of significant comorbidities, and ability to speak/read/understand English.

The multimodal lifestyle intervention has six foci: Positive cognition [mindset], Exercise/movement, Stress Reduction, Social Connection, Emotional Wellbeing, and Nutrition. All programming will take place online to maximize convenience/sustained participation.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older.
* Diagnosed with MGUS or SM based on commonly accepted criteria per the

International Multiple Myeloma Working Group (IMWG), defined as follows:

a. For a diagnosis of Smoldering Multiple Myeloma (SM), both criteria must be met: i. Serum monoclonal protein (IgG or IgA) ≥ 30g/L or urinary monoclonal protein ≥ 500mg per 24h and/or clonal bone marrow plasma cells 10-60% ii. Absence of myeloma-defining events or amyloidosis b. For a diagnosis of Non-IgM Monoclonal Gammopathy of Undetermined

Significance (MGUS):

i. Serum monoclonal protein <30g/L ii. Clonal bone marrow plasma cells <10% iii. Absence of end-organ damage such as hypercalcemia, renal insufficiency, anemia, and bone lesions (CRAB) or amyloidosis that can be attributed to the plasma cell proliferative disorder c. For a diagnosis of IgM MGUS: i. Serum IgM monoclonal protein <30g/L ii. No evidence of anemia, constitutional symptoms, hyperviscosity, lymphadenopathy, hepatosplenomegaly, or other end-organ damage that can be attributed to the plasma cell proliferative disorder d. For a diagnosis of light change MGUS: i. Abnormal FLC ratio (<0.26 or >1.65) ii. Increased level of the appropriate free light chain (increased κ FLC in patients with ratio >1.65 and increased λ FLC in patients with ratio <0.26) iii. No immunoglobulin heavy chain expression on immunofixation iv. Absence of end-organ damage such as hypercalcemia, renal insufficiency, anemia, and bone lesions (CRAB) or amyloidosis that can be attributed to the plasma cell proliferative disorder v. Clonal bone marrow plasma cells <10% vi. Urinary monoclonal protein <500mg/24h

* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2
* Ability to speak, read and comprehend the English language.
* Absence of significant intercurrent illness such as uncontrolled heart failure, unstable angina, cardiac arrhythmia and psychiatric illness which would preclude informed consent.
* Patient understands the purpose of the trial and procedures required for the trial, and can provide signed informed consent as which includes compliances with the requirements and restrictions listed in the informed consent form (ICF) and in the study protocol.
* Ability to adhere to the study visit schedule and all the protocol requirements, including surveillance imaging and test specimen (blood sample) collection at specified time points.

Exclusion Criteria:

* Evidence of any one or more of the following biomarkers of malignancy, or myeloma-defining events (MDEs) meeting IMWG criteria for a diagnosis of multiple myeloma:

  1. 60% or greater clonal plasma cells on bone marrow examination
  2. Serum involved / uninvolved free light chain ratio of 100 or greater, provided the absolute level of the involved light chain is at least 100mg/L (a patient's involved free light chain either kappa or lambda is the one that is above the normal reference range; the uninvolved free light chain is the one that is typically in, or below, the normal range)
  3. More than one focal lesion on MRI that is at least 5mm or greater in size.
* Evidence of end-organ damage as per the IMWG CRAB criteria, defined as follows:

  1. Hypercalcemia: serum calcium >0.25 mmol/L (>1mg/dL) higher than the upper limit of normal or >2.75 mmol/L (>11mg/dL)
  2. Renal insufficiency: creatinine clearance <40 mL per minute or serum creatinine >177mol/L (>2mg/dL)
  3. Anemia: hemoglobin value of >20g/L below the lowest limit of normal, or a hemoglobin value <100g/L
  4. Bone lesions: one or more osteolytic lesions on skeletal radiography, CT, or PET/CT. If bone marrow has <10% clonal plasma cells, more than one bone lesion is required to distinguish from solitary plasmacytoma with minimal marrow involvement
* Unwillingness or inability to follow required intervention behaviors, including any safety issues related to participating in any part of the intervention (e.g., a contraindication to gentle movement/exercise, BMI <18 kg/m2, etc.).
* Pregnancy or breastfeeding
* Patient has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the patient (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of multi-modal lifestyle intervention based on any of the 3 specified myeloma tumor burden biomarker surrogates | At study entry, 4 months, 8 months, and up to 12 months
  Efficacy of the multi-modal lifestyle intervention will be based on measurements of 3 myeloma-relevant biomarkers: M-Spike Protein, Free kappa light chains, and Free lambda-light chains. We will first determine which monoclonal protein is dominant for a given patient based on his/her/their individual lab values. These labs will be taken at baseline and compared to levels at 4-, 8-, and 12-month intervals to assess for changes in protein levels.

SECONDARY OUTCOMES:
Patient Acceptability (engagement) of the Lifestyle Intervention | At study entry, 4 months, 8 months, and up to 12 months
  Patient acceptability will be measured by a patient acceptability questionnaire
Patient Adherence (compliance) to the Lifestyle Intervention | At study entry, 4 months, 8 months, and up to 12 months
  Patient adherence will be measured based on attendance at clinic visits, the various scheduled individual and group meetings across all intervention components, and via the use of wearable technology

OTHER OUTCOMES:
Correlation between specified inflammation biomarkers and any of the 3 specified myeloma tumor burden biomarker surrogates | At study entry, 4 months, 8 months, and up to 12 months
  Inflammation will be measured using 3 surrogate markers: IL-6, TNF-alpha, and VEGF. These labs will be taken at baseline and compared to levels at 4-, 8-, and 12-month intervals to assess for a reduction in these levels and any observed correlation with myeloma markers
Correlation between patient glucose levels/changes and any of the 3 specified myeloma tumor burden biomarker surrogates | At study entry, 4 months, 8 months, and up to 12 months
  Fasting insulin levels and hemoglobin A1c (HbA1c) measurements will be taken at baseline and compared to levels at 4-, 8-, and 12-month intervals to assess for improvements and any observed correlation with designated myeloma markers. Average of In-Range Continuous Glucose Monitor (CGM) recordings will be calculated at baseline and compared to levels at 4-, 8-, and 12-month intervals to assess for improvements and correlation with select myeloma biomarkers.
Correlation between lipid-related biomarkers/changes and any of the 3 specified myeloma tumor burden biomarker surrogates | At study entry, 4 months, 8 months, and up to 12 months
  Body mass index (BMI), Abdominal Visceral Fat; High Density Lipoprotein - Cholesterol (HDL-C), Apolipoprotein A-1(APO A1), and Adiponectin will be measured at baseline and compared to levels at 4-, 8-, and 12-month intervals to assess for improvements and any correlation with the identified myeloma biomarkers
Validation of the PESSEN questionnaire | At study entry, 4 months, 8 months, and up to 12 months
  The PESSEN Questionnaire (Positive cognition, Emotional wellbeing, Social connection, Stress reduction, Exercise, Nutrition) is designed to assess a patient's overall lifestyle wellness as measured across six areas, assess the degree to which a patient believes that these six areas of lifestyle interventions can improve their cancer outcome, and to assign them a lifestyle wellness score.

CONTACTS AND LOCATIONS:
Overall Officials: David Siegel, MD, Principal Investigator — Hackensack Meridian Health

REFERENCES:
- [Background] Mateos MV, Landgren O. MGUS and Smoldering Multiple Myeloma: Diagnosis and Epidemiology. Cancer Treat Res. 2016;169:3-12. doi: 10.1007/978-3-319-40320-5_1. PMID 27696254
- [Background] Plano F, Corsale AM, Gigliotta E, Camarda G, Vullo C, Di Simone M, Shekarkar Azgomi M, Speciale M, Carlisi M, Caccamo N, Dieli F, Meraviglia S, Siragusa S, Botta C. Monoclonal Gammopathies and the Bone Marrow Microenvironment: From Bench to Bedside and Then Back Again. Hematol Rep. 2023 Jan 9;15(1):23-49. doi: 10.3390/hematolrep15010004. PMID 36648882
- [Background] Padala SA, Barsouk A, Barsouk A, Rawla P, Vakiti A, Kolhe R, Kota V, Ajebo GH. Epidemiology, Staging, and Management of Multiple Myeloma. Med Sci (Basel). 2021 Jan 20;9(1):3. doi: 10.3390/medsci9010003. PMID 33498356
- [Background] Cancer.Org. Published 2012. Https://Www.Cancer.Org/Cancer/Multiple-Myeloma/Detectiondiagnosis-Staging/Surviva l-Rates.Html. Accessed January 19, 2023.
- [Background] Multiple Myeloma - Statistics. Cancer.Net. Published February 28, 2019. Https://Www.Cancer.Net/Cancer-Types/Multiple-Myeloma/Statistics. Accessed January 19, 2023.
- [Background] Kyle RA, Remstein ED, Therneau TM, Dispenzieri A, Kurtin PJ, Hodnefield JM, Larson DR, Plevak MF, Jelinek DF, Fonseca R, Melton LJ 3rd, Rajkumar SV. Clinical course and prognosis of smoldering (asymptomatic) multiple myeloma. N Engl J Med. 2007 Jun 21;356(25):2582-90. doi: 10.1056/NEJMoa070389. PMID 17582068
- [Background] Mateos MV, Kumar S, Dimopoulos MA, Gonzalez-Calle V, Kastritis E, Hajek R, De Larrea CF, Morgan GJ, Merlini G, Goldschmidt H, Geraldes C, Gozzetti A, Kyriakou C, Garderet L, Hansson M, Zamagni E, Fantl D, Leleu X, Kim BS, Esteves G, Ludwig H, Usmani S, Min CK, Qi M, Ukropec J, Weiss BM, Rajkumar SV, Durie BGM, San-Miguel J. International Myeloma Working Group risk stratification model for smoldering multiple myeloma (SMM). Blood Cancer J. 2020 Oct 16;10(10):102. doi: 10.1038/s41408-020-00366-3. PMID 33067414
- [Background] Aljama MA, Sidiqi MH, Lakshman A, Dispenzieri A, Jevremovic D, Gertz MA, Lacy MQ, Buadi FK, Dingli D, Muchtar E, Fonder AL, Hayman SR, Hobbs MA, Gonsalves WI, Warsame R, Kourelis TV, Hwa YL, Kapoor P, Leung N, Go RS, Kyle RA, Rajkumar SV, Kumar SK. Plasma cell proliferative index is an independent predictor of progression in smoldering multiple myeloma. Blood Adv. 2018 Nov 27;2(22):3149-3154. doi: 10.1182/bloodadvances.2018024794. PMID 30463914
- [Background] Chang SH, Gumbel J, Luo S, Thomas TS, Sanfilippo KM, Luo J, Colditz GA, Carson KR. Post-MGUS Diagnosis Serum Monoclonal-Protein Velocity and the Progression of Monoclonal Gammopathy of Undetermined Significance to Multiple Myeloma. Cancer Epidemiol Biomarkers Prev. 2019 Dec;28(12):2055-2061. doi: 10.1158/1055-9965.EPI-19-0132. Epub 2019 Sep 9. PMID 31501149
- [Background] Shapiro YN, Peppercorn JM, Yee AJ, Branagan AR, Raje NS, Donnell EKO. Lifestyle considerations in multiple myeloma. Blood Cancer J. 2021 Oct 26;11(10):172. doi: 10.1038/s41408-021-00560-x. PMID 34702799
- [Background] Lee DH, Fung TT, Tabung FK, Marinac CR, Devore EE, Rosner BA, Ghobrial IM, Colditz GA, Giovannucci EL, Birmann BM. Prediagnosis dietary pattern and survival in patients with multiple myeloma. Int J Cancer. 2020 Oct 1;147(7):1823-1830. doi: 10.1002/ijc.32928. Epub 2020 Feb 28. PMID 32067221
- [Background] Lee DH, Fung TT, Tabung FK, Colditz GA, Ghobrial IM, Rosner BA, Giovannucci EL, Birmann BM. Dietary Pattern and Risk of Multiple Myeloma in Two Large Prospective US Cohort Studies. JNCI Cancer Spectr. 2019 Jun;3(2):pkz025. doi: 10.1093/jncics/pkz025. Epub 2019 Apr 27. PMID 31149654
- [Background] Aggarwal V, Kashyap D, Sak K, Tuli HS, Jain A, Chaudhary A, Garg VK, Sethi G, Yerer MB. Molecular Mechanisms of Action of Tocotrienols in Cancer: Recent Trends and Advancements. Int J Mol Sci. 2019 Feb 2;20(3):656. doi: 10.3390/ijms20030656. PMID 30717416
- [Background] Gong IY, Cheung MC, Read S, Na Y, Lega IC, Lipscombe LL. Association between diabetes and haematological malignancies: a population-based study. Diabetologia. 2021 Mar;64(3):540-551. doi: 10.1007/s00125-020-05338-7. Epub 2021 Jan 6. PMID 33409570
- [Background] Parikh R, Tariq SM, Marinac CR, Shah UA. A comprehensive review of the impact of obesity on plasma cell disorders. Leukemia. 2022 Feb;36(2):301-314. doi: 10.1038/s41375-021-01443-7. Epub 2021 Oct 15. PMID 34654885
- [Background] Hodge A, Sheean P, O'Connor P, Tyler K, Kerschner A, Williams A, Jensik K, Visotcky A, D'Souza A, Hari P, Dhakal B, Chhabra S, Flynn KE, Hagen P, Stolley M. Exploring health behaviors and the feasibility of a lifestyle intervention for patients with multiple myeloma. Support Care Cancer. 2022 Dec;30(12):9771-9779. doi: 10.1007/s00520-022-07385-9. Epub 2022 Oct 26. PMID 36287278
- [Background] Storti P, Agnelli L, Palma BD, Todoerti K, Marchica V, Accardi F, Sammarelli G, Deluca F, Toscani D, Costa F, Vicario E, Todaro G, Martella E, Neri A, Giuliani N. The transcriptomic profile of CD138+ cells from patients with early progression from smoldering to active multiple myeloma remains substantially unchanged. Haematologica. 2019 Oct;104(10):e465-e469. doi: 10.3324/haematol.2018.209999. Epub 2019 Mar 7. No abstract available. PMID 30846495
- [Background] Boyle EM, Deshpande S, Tytarenko R, Ashby C, Wang Y, Bauer MA, Johnson SK, Wardell CP, Thanendrarajan S, Zangari M, Facon T, Dumontet C, Barlogie B, Arbini A, Rustad EH, Maura F, Landgren O, Zhan F, van Rhee F, Schinke C, Davies FE, Morgan GJ, Walker BA. The molecular make up of smoldering myeloma highlights the evolutionary pathways leading to multiple myeloma. Nat Commun. 2021 Jan 12;12(1):293. doi: 10.1038/s41467-020-20524-2. PMID 33436579
- [Background] Madhira BR, Konala VM, Adapa S, Naramala S, Ravella PM, Parikh K, Gentile TC. Recent Advances in the Management of Smoldering Multiple Myeloma. World J Oncol. 2020 Apr;11(2):45-54. doi: 10.14740/wjon1245. Epub 2020 Mar 29. PMID 32284772
- [Background] Kim EB, Yee AJ, Raje N. Treatment of Smoldering Multiple Myeloma: Ready for Prime Time? Cancers (Basel). 2020 May 13;12(5):1223. doi: 10.3390/cancers12051223. PMID 32414145
- [Background] Romano A, Cerchione C, Conticello C, Martinelli G, Di Raimondo F. How we manage smoldering multiple myeloma. Hematol Rep. 2020 Sep 21;12(Suppl 1):8951. doi: 10.4081/hr.2020.8951. eCollection 2020 Sep 21. PMID 33042502
- [Background] San Miguel J, Mateos MV, Gonzalez V, et al. Updated risk stratification model for smoldering multiple myeloma (SMM) incorporating the revised IMWG diagnostic criteria. J Clin Oncol. 2019;37(15_suppl):8000-8000. doi:10.1200/JCO.2019.37.15_suppl.8000
- [Background] Ho M, Patel A, Goh CY, Moscvin M, Zhang L, Bianchi G. Changing paradigms in diagnosis and treatment of monoclonal gammopathy of undetermined significance (MGUS) and smoldering multiple myeloma (SMM). Leukemia. 2020 Dec;34(12):3111-3125. doi: 10.1038/s41375-020-01051-x. Epub 2020 Oct 12. PMID 33046818
- [Background] Boen CE, Barrow DA, Bensen JT, Farnan L, Gerstel A, Hendrix LH, Yang YC. Social Relationships, Inflammation, and Cancer Survival. Cancer Epidemiol Biomarkers Prev. 2018 May;27(5):541-549. doi: 10.1158/1055-9965.EPI-17-0836. Epub 2018 Feb 23. PMID 29475966
- [Background] Shah UA, Alicea D, Adintori PA, et al. A Pilot Plant-Based Dietary Intervention in Overweight and Obese Patients with Monoclonal Gammopathy of Undetermined Significance and Smoldering Multiple Myeloma- the Nutrition Prevention (NUTRIVENTION) Study. Blood. 2021;138(Supplement 1):4759-4759. doi:10.1182/blood-2021-151049
- [Background] Shah UA, Parikh R, Castro F, Bellone M, Lesokhin AM. Dietary and microbiome evidence in multiple myeloma and other plasma cell disorders. Leukemia. 2023 May;37(5):964-980. doi: 10.1038/s41375-023-01874-4. Epub 2023 Mar 30. PMID 36997677
- [Background] Shah UA, Maclachlan KH, Derkach A, Salcedo M, Barnett K, Caple J, Blaslov J, Tran L, Ciardiello A, Burge M, Shekarkhand T, Adintori P, Cross J, Pianko MJ, Hosszu K, McAvoy D, Mailankody S, Korde N, Hultcrantz M, Hassoun H, Tan CR, Lu SX, Patel D, Diamond B, Shah G, Scordo M, Lahoud O, Chung DJ, Landau H, Usmani SZ, Giralt S, Taur Y, Landgren CO, Block G, Block T, Peled JU, van den Brink MRM, Lesokhin AM. Sustained Minimal Residual Disease Negativity in Multiple Myeloma is Associated with Stool Butyrate and Healthier Plant-Based Diets. Clin Cancer Res. 2022 Dec 1;28(23):5149-5155. doi: 10.1158/1078-0432.CCR-22-0723. PMID 36170461
- [Background] Brevi A, Cogrossi LL, Lorenzoni M, Mattorre B, Bellone M. The Insider: Impact of the Gut Microbiota on Cancer Immunity and Response to Therapies in Multiple Myeloma. Front Immunol. 2022 Mar 17;13:845422. doi: 10.3389/fimmu.2022.845422. eCollection 2022. PMID 35371048
- [Background] Groeneveldt L, Mein G, Garrod R, Jewell AP, Van Someren K, Stephens R, D'Sa SP, Yong KL. A mixed exercise training programme is feasible and safe and may improve quality of life and muscle strength in multiple myeloma survivors. BMC Cancer. 2013 Jan 24;13:31. doi: 10.1186/1471-2407-13-31. PMID 23347597
- [Background] Jones LW, Eves ND, Waner E, Joy AA. Exercise therapy across the lung cancer continuum. Curr Oncol Rep. 2009 Jul;11(4):255-62. doi: 10.1007/s11912-009-0036-0. PMID 19508829
- [Background] Zheng A, Zhang L, Yang J, Yin X, Zhang T, Wu X, Ma X. Physical activity prevents tumor metastasis through modulation of immune function. Front Pharmacol. 2022 Oct 12;13:1034129. doi: 10.3389/fphar.2022.1034129. eCollection 2022. PMID 36313283
- [Background] Sitlinger A, Brander DM, Bartlett DB. Impact of exercise on the immune system and outcomes in hematologic malignancies. Blood Adv. 2020 Apr 28;4(8):1801-1811. doi: 10.1182/bloodadvances.2019001317. PMID 32343800
- [Background] Baldelli G, De Santi M, Gervasi M, Annibalini G, Sisti D, Hojman P, Sestili P, Stocchi V, Barbieri E, Brandi G. The effects of human sera conditioned by high-intensity exercise sessions and training on the tumorigenic potential of cancer cells. Clin Transl Oncol. 2021 Jan;23(1):22-34. doi: 10.1007/s12094-020-02388-6. Epub 2020 May 23. PMID 32447643
- [Background] Sitlinger A, Deal MA, Garcia E, Connelly M, Thompson D, Stewart T, Macdonald G, Hanson ED, Neely M, Neely B, Artese A, Weinberg JB, Brander D, Bartlett DB. Associations of clinical and circulating metabolic biomarkers with low physical fitness and function in adults with chronic lymphocytic leukemia. Front Oncol. 2022 Aug 3;12:933619. doi: 10.3389/fonc.2022.933619. eCollection 2022. PMID 35992862
- [Background] Wang J, Sheng L, Lai Y, Ouyang G, Xu Z. Effects of physical activity on clinical and inflammatory markers in diagnosing multiple myeloma patients. Front Physiol. 2023 Jan 4;13:1094470. doi: 10.3389/fphys.2022.1094470. eCollection 2022. PMID 36685193
- [Background] Lecat CSY, McCourt O, Land J, Yong K, Fisher A. Multiple myeloma and physical activity. BMC Res Notes. 2021 May 7;14(1):171. doi: 10.1186/s13104-021-05591-y. PMID 33962674
- [Background] Hillengass M, Joseph J, Mccarthy J, Hillengass J. Physical Activity in Multiple Myeloma: A Review of the Current Literature. J Adv Pract Oncol. 2023 Mar;14(2):153-158. doi: 10.6004/jadpro.2023.14.2.5. Epub 2023 Mar 1. PMID 37009406
- [Background] Joseph JM, Hillengass M, Jacobson H, et al. Immune Markers of Multiple Myeloma Patients Demonstrate Significant Change after Participation in Six-Month Physical Activity Intervention. Blood. 2022;140(Supplement 1):12630-12632. doi:10.1182/blood-2022-167655
- [Background] Roswell Park Cancer Institute. Strength Training in Improving Pain and Quality of Life in Patients With Multiple Myeloma. ClinicalTrials.Gov Identifier: NCT03793907. Updated April 10, 2023. Accessed May 19, 2023. Https://Clinicaltrials.Gov/Ct2/Show/NCT03793907
- [Background] Hillengass J, Hillengass M, Sweeney NW, et al. Physical Activity in Patients with Monoclonal Gammopathies - a Healthtree Cure Hub Study. Blood. 2022;140(Supplement 1):7136-7137. doi:10.1182/blood-2022-162327
- [Background] Seefried L, Genest F, Stromsdorfer J, Engelmann B, Lapa C, Jakob F, Baumann FT, Sperlich B, Jundt F. Impact of whole-body vibration exercise on physical performance and bone turnover in patients with monoclonal gammopathy of undetermined significance. J Bone Oncol. 2020 Sep 28;25:100323. doi: 10.1016/j.jbo.2020.100323. eCollection 2020 Dec. PMID 33083217
- [Background] Strasser F, Palmer JL, Schover LR, Yusuf SW, Pisters K, Vassilopoulou-Sellin R, DeGracia B, Willey JS, Bruera E. The impact of hypogonadism and autonomic dysfunction on fatigue, emotional function, and sexual desire in male patients with advanced cancer: a pilot study. Cancer. 2006 Dec 15;107(12):2949-57. doi: 10.1002/cncr.22339. PMID 17103445
- [Background] Walsh D, Nelson KA. Autonomic nervous system dysfunction in advanced cancer. Support Care Cancer. 2002 Oct;10(7):523-8. doi: 10.1007/s00520-002-0376-x. Epub 2002 Aug 22. PMID 12324806
- [Background] Magnon C, Hall SJ, Lin J, Xue X, Gerber L, Freedland SJ, Frenette PS. Autonomic nerve development contributes to prostate cancer progression. Science. 2013 Jul 12;341(6142):1236361. doi: 10.1126/science.1236361. PMID 23846904
- [Background] De Couck M, Caers R, Spiegel D, Gidron Y. The Role of the Vagus Nerve in Cancer Prognosis: A Systematic and a Comprehensive Review. J Oncol. 2018 Jul 2;2018:1236787. doi: 10.1155/2018/1236787. eCollection 2018. PMID 30057605
- [Background] Yang EV. Role for catecholamines in tumor progression: possible use for beta-blockers in the treatment of cancer. Cancer Biol Ther. 2010 Jul 1;10(1):30-2. doi: 10.4161/cbt.10.1.12260. Epub 2010 Jul 6. No abstract available. PMID 20505322
- [Background] Hanns P, Paczulla AM, Medinger M, Konantz M, Lengerke C. Stress and catecholamines modulate the bone marrow microenvironment to promote tumorigenesis. Cell Stress. 2019 Jun 4;3(7):221-235. doi: 10.15698/cst2019.07.192. PMID 31338489
- [Background] Yang EV, Benson DM, Glaser R. Catecholamines can mediate stress-related effects on tumor progression. Expert Rev Endocrinol Metab. 2008 Nov;3(6):699-703. doi: 10.1586/17446651.3.6.699. PMID 30764060
- [Background] Zhou X, Ma Z, Zhang L, Zhou S, Wang J, Wang B, Fu W. Heart rate variability in the prediction of survival in patients with cancer: A systematic review and meta-analysis. J Psychosom Res. 2016 Oct;89:20-5. doi: 10.1016/j.jpsychores.2016.08.004. Epub 2016 Aug 8. PMID 27663106
- [Background] Hanoun M, Maryanovich M, Arnal-Estape A, Frenette PS. Neural regulation of hematopoiesis, inflammation, and cancer. Neuron. 2015 Apr 22;86(2):360-73. doi: 10.1016/j.neuron.2015.01.026. PMID 25905810
- [Background] Cheng Y, Sun F, D'Souza A, Dhakal B, Pisano M, Chhabra S, Stolley M, Hari P, Janz S. Autonomic nervous system control of multiple myeloma. Blood Rev. 2021 Mar;46:100741. doi: 10.1016/j.blre.2020.100741. Epub 2020 Aug 11. PMID 32807576
- [Background] Zhang L, Pan J, Chen W, Jiang J, Huang J. Chronic stress-induced immune dysregulation in cancer: implications for initiation, progression, metastasis, and treatment. Am J Cancer Res. 2020 May 1;10(5):1294-1307. eCollection 2020. PMID 32509380
- [Background] Finkelstein-Fox L, Denninger JW, Walsh LE, Laubach JP, Yee AJ, O'Donnell E, Macklin EA, Gu X, Muzikansky A, Libermann TA, Nicolosi G, Richardson PG, Raje NS, Fricchione GL, Perez GK, Traeger LN, Chad-Friedman E, Park ER. Psychosocial and NF-kappaB Activity Effects of the Stress Management and Resiliency Training: Relaxation Response Resiliency Program (SMART-3RP) on Patients With MGUS and Smoldering Multiple Myeloma: A Randomized Waitlist Control Trial. Psychooncology. 2025 Jul;34(7):e70216. doi: 10.1002/pon.70216. PMID 40681960
- [Background] Maatouk I, He S, Hummel M, Hemmer S, Hillengass M, Goldschmidt H, Hartmann M, Herzog W, Hillengass J. Patients with precursor disease exhibit similar psychological distress and mental HRQOL as patients with active myeloma. Blood Cancer J. 2019 Jan 21;9(2):9. doi: 10.1038/s41408-019-0172-1. No abstract available. PMID 30664623
- [Background] Wang YH, Li JQ, Shi JF, Que JY, Liu JJ, Lappin JM, Leung J, Ravindran AV, Chen WQ, Qiao YL, Shi J, Lu L, Bao YP. Depression and anxiety in relation to cancer incidence and mortality: a systematic review and meta-analysis of cohort studies. Mol Psychiatry. 2020 Jul;25(7):1487-1499. doi: 10.1038/s41380-019-0595-x. Epub 2019 Nov 19. PMID 31745237
- [Background] Maatouk I, He S, Becker N, Hummel M, Hemmer S, Hillengass M, Goldschmidt H, Hartmann M, Schellberg D, Herzog W, Hillengass J. Association of resilience with health-related quality of life and depression in multiple myeloma and its precursors: results of a German cross-sectional study. BMJ Open. 2018 Jul 30;8(7):e021376. doi: 10.1136/bmjopen-2017-021376. PMID 30061438
- [Background] Kroenke CH, Michael YL, Poole EM, Kwan ML, Nechuta S, Leas E, Caan BJ, Pierce J, Shu XO, Zheng Y, Chen WY. Postdiagnosis social networks and breast cancer mortality in the After Breast Cancer Pooling Project. Cancer. 2017 Apr 1;123(7):1228-1237. doi: 10.1002/cncr.30440. Epub 2016 Dec 12. PMID 27943274
- [Background] Terao T, Tsushima T, Miura D, Narita K, Takeuchi M, Matsue K. Social frailty predicts worse outcomes in patients with multiple myeloma: A novelty in an old approach. EJHaem. 2020 Jun 17;1(1):103-112. doi: 10.1002/jha2.40. eCollection 2020 Jul. PMID 35847687
- [Background] Seyfried TN, Flores RE, Poff AM, D'Agostino DP. Cancer as a metabolic disease: implications for novel therapeutics. Carcinogenesis. 2014 Mar;35(3):515-27. doi: 10.1093/carcin/bgt480. Epub 2013 Dec 16. PMID 24343361
- [Background] Le A, Udupa S, Zhang C. The Metabolic Interplay between Cancer and Other Diseases. Trends Cancer. 2019 Dec;5(12):809-821. doi: 10.1016/j.trecan.2019.10.012. Epub 2019 Nov 21. PMID 31813458
- [Background] Ragbourne SC, Maghsoodi N, Streetly M, Crook MA. The Association between Metabolic Syndrome and Multiple Myeloma. Acta Haematol. 2021;144(1):24-33. doi: 10.1159/000505992. Epub 2020 May 14. PMID 32408305
- [Background] Gavriatopoulou M, Paschou SA, Ntanasis-Stathopoulos I, Dimopoulos MA. Metabolic Disorders in Multiple Myeloma. Int J Mol Sci. 2021 Oct 22;22(21):11430. doi: 10.3390/ijms222111430. PMID 34768861
- [Background] Georgakopoulou R, Andrikopoulou A, Sergentanis TN, Fiste O, Zagouri F, Gavriatopoulou M, Psaltopoulou T, Kastritis E, Terpos E, Dimopoulos MA. Overweight/Obesity and Monoclonal Gammopathy of Undetermined Significance. Clin Lymphoma Myeloma Leuk. 2021 Jun;21(6):361-367. doi: 10.1016/j.clml.2021.01.008. Epub 2021 Jan 15. PMID 33582053
- [Background] Chang SH, Luo S, Thomas TS, O'Brian KK, Colditz GA, Carlsson NP, Carson KR. Obesity and the Transformation of Monoclonal Gammopathy of Undetermined Significance to Multiple Myeloma: A Population-Based Cohort Study. J Natl Cancer Inst. 2016 Dec 31;109(5):djw264. doi: 10.1093/jnci/djw264. Print 2017 May. PMID 28040690
- [Background] Markus E, Trestman S, Cohen Y, Angel Y, Sofer Y, Mittelman M, Avivi I, Stern N, Izkhakov E. Components of metabolic syndrome in patients with multiple myeloma and smoldering multiple myeloma. BMC Cancer. 2020 May 30;20(1):489. doi: 10.1186/s12885-020-06976-1. PMID 32473631
- [Background] Morris EV, Edwards CM. Adipokines, adiposity, and bone marrow adipocytes: Dangerous accomplices in multiple myeloma. J Cell Physiol. 2018 Dec;233(12):9159-9166. doi: 10.1002/jcp.26884. Epub 2018 Jun 26. PMID 29943829
- [Background] Shen Y, Wang C, Wang Y, Lu J, Chen L, Zhang L, Lu W, Zhu W, Hu G, Xia T, Zhou J. Association between time in range and cancer mortality among patients with type 2 diabetes: a prospective cohort study. Chin Med J (Engl). 2021 Sep 15;135(3):288-294. doi: 10.1097/CM9.0000000000001740. PMID 34995040
- [Background] Gabbay MAL, Rodacki M, Calliari LE, Vianna AGD, Krakauer M, Pinto MS, Reis JS, Punales M, Miranda LG, Ramalho AC, Franco DR, Pedrosa HPC. Time in range: a new parameter to evaluate blood glucose control in patients with diabetes. Diabetol Metab Syndr. 2020 Mar 16;12:22. doi: 10.1186/s13098-020-00529-z. eCollection 2020. PMID 32190124
- [Background] Golombick T, Diamond TH, Manoharan A, Ramakrishna R. Monoclonal gammopathy of undetermined significance, smoldering multiple myeloma, and curcumin: a randomized, double-blind placebo-controlled cross-over 4g study and an open-label 8g extension study. Am J Hematol. 2012 May;87(5):455-60. doi: 10.1002/ajh.23159. Epub 2012 Apr 4. PMID 22473809
- [Background] Golombick T, Diamond TH, Badmaev V, Manoharan A, Ramakrishna R. The potential role of curcumin in patients with monoclonal gammopathy of undefined significance--its effect on paraproteinemia and the urinary N-telopeptide of type I collagen bone turnover marker. Clin Cancer Res. 2009 Sep 15;15(18):5917-22. doi: 10.1158/1078-0432.CCR-08-2217. Epub 2009 Sep 8. PMID 19737963
- [Background] Mirzaei H, Bagheri H, Ghasemi F, Khoi JM, Pourhanifeh MH, Heyden YV, Mortezapour E, Nikdasti A, Jeandet P, Khan H, Sahebkar A. Anti-Cancer Activity of Curcumin on Multiple Myeloma. Anticancer Agents Med Chem. 2021;21(5):575-586. doi: 10.2174/1871520620666200918113625. PMID 32951583
- [Background] Deguchi A. Curcumin targets in inflammation and cancer. Endocr Metab Immune Disord Drug Targets. 2015;15(2):88-96. doi: 10.2174/1871530315666150316120458. PMID 25772169
- [Background] Santosa D, Suharti C, Riwanto I, Dharmana E, Pangarsa EA, Setiawan B, Suyono S, Tobing ML, Suhartono S, Hadisapurto S. Curcumin as adjuvant therapy to improve remission in myeloma patients: A pilot randomized clinical trial. Caspian J Intern Med. 2022 Spring;13(2):375-384. doi: 10.22088/cjim.13.2.9. PMID 35919637
- [Background] Zhan F, Barlogie B, Arzoumanian V, Huang Y, Williams DR, Hollmig K, Pineda-Roman M, Tricot G, van Rhee F, Zangari M, Dhodapkar M, Shaughnessy JD Jr. Gene-expression signature of benign monoclonal gammopathy evident in multiple myeloma is linked to good prognosis. Blood. 2007 Feb 15;109(4):1692-700. doi: 10.1182/blood-2006-07-037077. Epub 2006 Oct 5. PMID 17023574
- [Background] Kierkegaard-Brøchner S, Sørensen UM, Lange LB, Mortensen LS, Bruun JM. The outcome of a multicomponent lifestyle intervention in patients with obesity: A cohort study. Eur J IntegrMed. 2023;60:102259. doi:10.1016/j.eujim.2023.102259
- [Background] Wong VW, Ho FY, Shi NK, Sarris J, Chung KF, Yeung WF. Lifestyle medicine for depression: A meta-analysis of randomized controlled trials. J Affect Disord. 2021 Apr 1;284:203-216. doi: 10.1016/j.jad.2021.02.012. Epub 2021 Feb 5. PMID 33609955
- [Background] Wong VW, Ho FY, Shi NK, Sarris J, Ng CH, Tam OK. Lifestyle medicine for anxiety symptoms: A meta-analysis of randomized controlled trials. J Affect Disord. 2022 Aug 1;310:354-368. doi: 10.1016/j.jad.2022.04.151. Epub 2022 May 3. PMID 35523299
- [Background] Abbott S, Smith E, Tighe B, Lycett D. Group versus one-to-one multi-component lifestyle interventions for weight management: a systematic review and meta-analysis of randomised controlled trials. J Hum Nutr Diet. 2021 Jun;34(3):485-493. doi: 10.1111/jhn.12853. Epub 2020 Dec 28. PMID 33368624
- [Background] van Namen M, Prendergast L, Peiris C. Supervised lifestyle intervention for people with metabolic syndrome improves outcomes and reduces individual risk factors of metabolic syndrome: A systematic review and meta-analysis. Metabolism. 2019 Dec;101:153988. doi: 10.1016/j.metabol.2019.153988. Epub 2019 Oct 28. PMID 31672441
- [Background] Elvsaas IKO, Giske L, Fure B, Juvet LK. Multicomponent Lifestyle Interventions for Treating Overweight and Obesity in Children and Adolescents: A Systematic Review and Meta-Analyses. J Obes. 2017;2017:5021902. doi: 10.1155/2017/5021902. Epub 2017 Dec 17. PMID 29391949
- [Background] Petrogianni M, Kanellakis S, Kallianioti K, Argyropoulou D, Pitsavos C, Manios Y. A multicomponent lifestyle intervention produces favourable changes in diet quality and cardiometabolic risk indices in hypercholesterolaemic adults. J Hum Nutr Diet. 2013 Dec;26(6):596-605. doi: 10.1111/jhn.12041. Epub 2013 Mar 20. PMID 23510154
- [Background] Goyer L, Dufour R, Janelle C, Blais C, L'Abbe C, Raymond E, de Champlain J, Larochelle P. Randomized controlled trial on the long-term efficacy of a multifaceted, interdisciplinary lifestyle intervention in reducing cardiovascular risk and improving lifestyle in patients at risk of cardiovascular disease. J Behav Med. 2013 Apr;36(2):212-24. doi: 10.1007/s10865-012-9407-3. Epub 2012 Mar 9. PMID 22402823
- [Background] Golubic M, Schneeberger D, Kirkpatrick K, Bar J, Bernstein A, Weems F, Ehrman J, Perko J, Doyle J, Roizen M. Comprehensive Lifestyle Modification Intervention to Improve Chronic Disease Risk Factors and Quality of Life in Cancer Survivors. J Altern Complement Med. 2018 Nov;24(11):1085-1091. doi: 10.1089/acm.2018.0193. Epub 2018 Aug 1. PMID 30067063
- [Background] Ricanati EH, Golubic M, Yang D, Saager L, Mascha EJ, Roizen MF. Mitigating preventable chronic disease: Progress report of the Cleveland Clinic's Lifestyle 180 program. Nutr Metab (Lond). 2011 Nov 23;8:83. doi: 10.1186/1743-7075-8-83. PMID 22112436
- [Background] Innao V, Allegra A, Ginaldi L, Pioggia G, De Martinis M, Musolino C, Gangemi S. Reviewing the Significance of Vitamin D Substitution in Monoclonal Gammopathies. Int J Mol Sci. 2021 May 6;22(9):4922. doi: 10.3390/ijms22094922. PMID 34066482
- [Background] Gile JJ, Lopez CL, Ruan GJ, Hathcock MA, Abeykoon JP, Heimgartner JR, Baumann NA, McMahon MM, Micallef IN, Johnston PB, Bisneto JCV, Porrata LF, Paludo J, Ansell SM, Hogan WJ, Witzig TE. Hypomagnesemia at the time of autologous stem cell transplantation for patients with diffuse large B-cell lymphoma is associated with an increased risk of failure. Blood Cancer J. 2021 Mar 26;11(3):65. doi: 10.1038/s41408-021-00452-0. PMID 33771971
- [Background] Bharti AC, Donato N, Singh S, Aggarwal BB. Curcumin (diferuloylmethane) down-regulates the constitutive activation of nuclear factor-kappa B and IkappaBalpha kinase in human multiple myeloma cells, leading to suppression of proliferation and induction of apoptosis. Blood. 2003 Feb 1;101(3):1053-62. doi: 10.1182/blood-2002-05-1320. Epub 2002 Sep 5. PMID 12393461
- [Background] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. BMJ. 2021 Sep 30;374:n2061. doi: 10.1136/bmj.n2061. PMID 34593508
- [Background] Klaic M, Kapp S, Hudson P, Chapman W, Denehy L, Story D, Francis JJ. Implementability of healthcare interventions: an overview of reviews and development of a conceptual framework. Implement Sci. 2022 Jan 27;17(1):10. doi: 10.1186/s13012-021-01171-7. PMID 35086538
- [Background] Paynter C, McDonald C, Story D, Francis JJ. Application of the theoretical framework of acceptability in a surgical setting: Theoretical and methodological insights. Br J Health Psychol. 2023 Nov;28(4):1153-1168. doi: 10.1111/bjhp.12677. Epub 2023 Jun 24. PMID 37353989
- [Background] Coleman EA, Coon S, Hall-Barrow J, Richards K, Gaylor D, Stewart B. Feasibility of exercise during treatment for multiple myeloma. Cancer Nurs. 2003 Oct;26(5):410-9. doi: 10.1097/00002820-200310000-00012. PMID 14710804
- [Background] Larsen RF, Jarden M, Minet LR, Frolund UC, Abildgaard N. Supervised and home-based physical exercise in patients newly diagnosed with multiple myeloma-a randomized controlled feasibility study. Pilot Feasibility Stud. 2019 Nov 12;5:130. doi: 10.1186/s40814-019-0518-2. eCollection 2019. PMID 31741745
- [Background] Lavery JA, Boutros PC, Knight D, Tammela T, Moskowitz CS, Jones LW. Association of exercise with pan-cancer incidence and overall survival. Cancer Cell. 2024 Feb 12;42(2):169-171. doi: 10.1016/j.ccell.2023.12.007. Epub 2024 Jan 4. PMID 38181796
- [Background] Coleman EA, Coon SK, Kennedy RL, Lockhart KD, Stewart CB, Anaissie EJ, Barlogie B. Effects of exercise in combination with epoetin alfa during high-dose chemotherapy and autologous peripheral blood stem cell transplantation for multiple myeloma. Oncol Nurs Forum. 2008 May;35(3):E53-61. doi: 10.1188/08.ONF.E53-E61. PMID 18467280
- [Background] Sheinboim D, Parikh S, Manich P, Markus I, Dahan S, Parikh R, Stubbs E, Cohen G, Zemser-Werner V, Bell RE, Ruiz SA, Percik R, Brenner R, Leibou S, Vaknine H, Arad G, Gerber Y, Keinan-Boker L, Shimony T, Bikovski L, Goldstein N, Constantini K, Labes S, Mordechai S, Doron H, Lonescu A, Ziv T, Nizri E, Choshen G, Eldar-Finkelman H, Tabach Y, Helman A, Ben-Eliyahu S, Erez N, Perlson E, Geiger T, Ben-Zvi D, Khaled M, Gepner Y, Levy C. An Exercise-Induced Metabolic Shield in Distant Organs Blocks Cancer Progression and Metastatic Dissemination. Cancer Res. 2022 Nov 15;82(22):4164-4178. doi: 10.1158/0008-5472.CAN-22-0237. PMID 36084256
- [Background] Zheng G, Qiu P, Xia R, Lin H, Ye B, Tao J, Chen L. Effect of Aerobic Exercise on Inflammatory Markers in Healthy Middle-Aged and Older Adults: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Front Aging Neurosci. 2019 Apr 26;11:98. doi: 10.3389/fnagi.2019.00098. eCollection 2019. PMID 31080412
- [Background] Dimitrov S, Hulteng E, Hong S. Inflammation and exercise: Inhibition of monocytic intracellular TNF production by acute exercise via beta2-adrenergic activation. Brain Behav Immun. 2017 Mar;61:60-68. doi: 10.1016/j.bbi.2016.12.017. Epub 2016 Dec 21. PMID 28011264
- [Background] Gleeson M, Bishop NC, Stensel DJ, Lindley MR, Mastana SS, Nimmo MA. The anti-inflammatory effects of exercise: mechanisms and implications for the prevention and treatment of disease. Nat Rev Immunol. 2011 Aug 5;11(9):607-15. doi: 10.1038/nri3041. PMID 21818123
- [Background] Nery C, Moraes SRA, Novaes KA, Bezerra MA, Silveira PVC, Lemos A. Effectiveness of resistance exercise compared to aerobic exercise without insulin therapy in patients with type 2 diabetes mellitus: a meta-analysis. Braz J Phys Ther. 2017 Nov-Dec;21(6):400-415. doi: 10.1016/j.bjpt.2017.06.004. Epub 2017 Jul 5. PMID 28728958
- [Background] Magkos F, Tsekouras Y, Kavouras SA, Mittendorfer B, Sidossis LS. Improved insulin sensitivity after a single bout of exercise is curvilinearly related to exercise energy expenditure. Clin Sci (Lond). 2008 Jan;114(1):59-64. doi: 10.1042/CS20070134. PMID 17635103
- [Background] Franczyk B, Gluba-Brzozka A, Cialkowska-Rysz A, Lawinski J, Rysz J. The Impact of Aerobic Exercise on HDL Quantity and Quality: A Narrative Review. Int J Mol Sci. 2023 Feb 28;24(5):4653. doi: 10.3390/ijms24054653. PMID 36902082
- [Background] Becic T, Studenik C, Hoffmann G. Exercise Increases Adiponectin and Reduces Leptin Levels in Prediabetic and Diabetic Individuals: Systematic Review and Meta-Analysis of Randomized Controlled Trials. Med Sci (Basel). 2018 Oct 30;6(4):97. doi: 10.3390/medsci6040097. PMID 30380802
- [Background] Wang Y, Shen L, Xu D. Aerobic exercise reduces triglycerides by targeting apolipoprotein C3 in patients with coronary heart disease. Clin Cardiol. 2019 Jan;42(1):56-61. doi: 10.1002/clc.23104. Epub 2018 Dec 21. PMID 30511426
- [Background] Momma H, Kawakami R, Honda T, Sawada SS. Muscle-strengthening activities are associated with lower risk and mortality in major non-communicable diseases: a systematic review and meta-analysis of cohort studies. Br J Sports Med. 2022 Jul;56(13):755-763. doi: 10.1136/bjsports-2021-105061. Epub 2022 Feb 28. PMID 35228201
- [Background] Nascimento W, Ferrari G, Martins CB, Rey-Lopez JP, Izquierdo M, Lee DH, Giovannucci EL, Rezende LFM. Muscle-strengthening activities and cancer incidence and mortality: a systematic review and meta-analysis of observational studies. Int J Behav Nutr Phys Act. 2021 May 29;18(1):69. doi: 10.1186/s12966-021-01142-7. PMID 34051796
- [Background] Parra-Soto S, Pell JP, Celis-Morales C, Ho FK. Absolute and relative grip strength as predictors of cancer: prospective cohort study of 445 552 participants in UK Biobank. J Cachexia Sarcopenia Muscle. 2022 Feb;13(1):325-332. doi: 10.1002/jcsm.12863. Epub 2021 Dec 24. PMID 34953058
- [Background] Massy-Westropp NM, Gill TK, Taylor AW, Bohannon RW, Hill CL. Hand Grip Strength: age and gender stratified normative data in a population-based study. BMC Res Notes. 2011 Apr 14;4:127. doi: 10.1186/1756-0500-4-127. PMID 21492469
- [Background] Cristian A. The sit to stand test in cancer patients and survivors. J Clin Oncol. 2023;41(16_suppl):e24058-e24058. doi:10.1200/JCO.2023.41.16_suppl.e24058
- [Background] Cristian A, Rubens M, Cristian C, Wang G, Mendez J. Characterization of Physical Function and Cancer-Related Physical Impairments in Hispanic Women With Breast Cancer: A Descriptive Study. Hisp Health Care Int. 2023 Dec;21(4):195-202. doi: 10.1177/15404153231183447. Epub 2023 Jun 20. PMID 37340714
- [Background] Brouha L. The Step Test: A Simple Method of Measuring Physical Fitness for Muscular Work in Young Men. Res Q Am Assoc Health Phys Educ Recreat. 1943;14(1):31-37. doi:10.1080/10671188.1943.10621204
- [Background] White KR, Lu J, Ibrahim Z, Furth PA. Enabling exercise prescription for survivors of cancer. Sci Rep. 2021 May 5;11(1):9557. doi: 10.1038/s41598-021-89021-w. PMID 33953311
- [Background] Kang SJ, Ha GC, Ko KJ. Association between resting heart rate, metabolic syndrome and cardiorespiratory fitness in Korean male adults. J Exerc Sci Fit. 2017 Jun;15(1):27-31. doi: 10.1016/j.jesf.2017.06.001. Epub 2017 Jun 20. PMID 29541128
- [Background] Jiang X, Liu X, Wu S, Zhang GQ, Peng M, Wu Y, Zheng X, Ruan C, Zhang W. Metabolic syndrome is associated with and predicted by resting heart rate: a cross-sectional and longitudinal study. Heart. 2015 Jan;101(1):44-9. doi: 10.1136/heartjnl-2014-305685. Epub 2014 Sep 1. PMID 25179964
- [Background] Rogowski O, Steinvil A, Berliner S, Cohen M, Saar N, Ben-Bassat OK, Shapira I. Elevated resting heart rate is associated with the metabolic syndrome. Cardiovasc Diabetol. 2009 Oct 14;8:55. doi: 10.1186/1475-2840-8-55. PMID 19828043
- [Background] Gutierrez-Martinez L, Brellenthin AG, Lefferts EC, Lee DC, Sui X, Lavie CJ, Blair SN. Resting Heart Rate and Risk of Cancer Mortality. Cancer Epidemiol Biomarkers Prev. 2021 Jun;30(6):1072-1078. doi: 10.1158/1055-9965.EPI-20-1731. Epub 2021 Apr 7. PMID 33827985
- [Background] Saint-Maurice PF, Troiano RP, Bassett DR Jr, Graubard BI, Carlson SA, Shiroma EJ, Fulton JE, Matthews CE. Association of Daily Step Count and Step Intensity With Mortality Among US Adults. JAMA. 2020 Mar 24;323(12):1151-1160. doi: 10.1001/jama.2020.1382. PMID 32207799
- [Background] Paluch AE, Bajpai S, Bassett DR, Carnethon MR, Ekelund U, Evenson KR, Galuska DA, Jefferis BJ, Kraus WE, Lee IM, Matthews CE, Omura JD, Patel AV, Pieper CF, Rees-Punia E, Dallmeier D, Klenk J, Whincup PH, Dooley EE, Pettee Gabriel K, Palta P, Pompeii LA, Chernofsky A, Larson MG, Vasan RS, Spartano N, Ballin M, Nordstrom P, Nordstrom A, Anderssen SA, Hansen BH, Cochrane JA, Dwyer T, Wang J, Ferrucci L, Liu F, Schrack J, Urbanek J, Saint-Maurice PF, Yamamoto N, Yoshitake Y, Newton RL Jr, Yang S, Shiroma EJ, Fulton JE; Steps for Health Collaborative. Daily steps and all-cause mortality: a meta-analysis of 15 international cohorts. Lancet Public Health. 2022 Mar;7(3):e219-e228. doi: 10.1016/S2468-2667(21)00302-9. PMID 35247352
- [Background] Vignjevic Petrinovic S, Milosevic MS, Markovic D, Momcilovic S. Interplay between stress and cancer-A focus on inflammation. Front Physiol. 2023 Mar 20;14:1119095. doi: 10.3389/fphys.2023.1119095. eCollection 2023. PMID 37020461
- [Background] Dhabhar FS. Effects of stress on immune function: the good, the bad, and the beautiful. Immunol Res. 2014 May;58(2-3):193-210. doi: 10.1007/s12026-014-8517-0. PMID 24798553
- [Background] Bosseboeuf A, Allain-Maillet S, Mennesson N, Tallet A, Rossi C, Garderet L, Caillot D, Moreau P, Piver E, Girodon F, Perreault H, Brouard S, Nicot A, Bigot-Corbel E, Hermouet S, Harb J. Pro-inflammatory State in Monoclonal Gammopathy of Undetermined Significance and in Multiple Myeloma Is Characterized by Low Sialylation of Pathogen-Specific and Other Monoclonal Immunoglobulins. Front Immunol. 2017 Oct 19;8:1347. doi: 10.3389/fimmu.2017.01347. eCollection 2017. PMID 29098000
- [Background] Nair S, Sng J, Boddupalli CS, Seckinger A, Chesi M, Fulciniti M, Zhang L, Rauniyar N, Lopez M, Neparidze N, Parker T, Munshi NC, Sexton R, Barlogie B, Orlowski R, Bergsagel L, Hose D, Flavell RA, Mistry PK, Meffre E, Dhodapkar MV. Antigen-mediated regulation in monoclonal gammopathies and myeloma. JCI Insight. 2018 Apr 19;3(8):e98259. doi: 10.1172/jci.insight.98259. eCollection 2018 Apr 19. PMID 29669929
- [Background] Mitchell AM, Crane PA, Kim Y. Perceived stress in survivors of suicide: psychometric properties of the Perceived Stress Scale. Res Nurs Health. 2008 Dec;31(6):576-85. doi: 10.1002/nur.20284. PMID 18449942
- [Background] Roberti JW, Harrington LN, Storch EA. Further Psychometric Support for the 10-Item Version of the Perceived Stress Scale. J Coll Couns. 2006;9(2):135-147. doi:10.1002/j.2161-1882.2006.tb00100.x
- [Background] Wu SM, Amtmann D. Psychometric Evaluation of the Perceived Stress Scale in Multiple Sclerosis. ISRN Rehabil. 2013;2013:1-9. doi:10.1155/2013/608356
- [Background] Kloter E, Barrueto K, Klein SD, Scholkmann F, Wolf U. Heart Rate Variability as a Prognostic Factor for Cancer Survival - A Systematic Review. Front Physiol. 2018 May 29;9:623. doi: 10.3389/fphys.2018.00623. eCollection 2018. PMID 29896113
- [Background] Tegegne BS, Man T, van Roon AM, Snieder H, Riese H. Reference values of heart rate variability from 10-second resting electrocardiograms: the Lifelines Cohort Study. Eur J Prev Cardiol. 2020 Dec;27(19):2191-2194. doi: 10.1177/2047487319872567. Epub 2019 Sep 9. No abstract available. PMID 31500461
- [Background] Holt-Lunstad J. Loneliness and Social Isolation as Risk Factors: The Power of Social Connection in Prevention. Am J Lifestyle Med. 2021 May 6;15(5):567-573. doi: 10.1177/15598276211009454. eCollection 2021 Sep-Oct. PMID 34646109
- [Background] Lubben JE. Assessing social networks among elderly populations: Fam Community Health. 1988;11(3):42-52. doi:10.1097/00003727-198811000-00008
- [Background] Yang M, Zhang Z, Nice EC, Wang C, Zhang W, Huang C. Psychological intervention to treat distress: An emerging frontier in cancer prevention and therapy. Biochim Biophys Acta Rev Cancer. 2022 Jan;1877(1):188665. doi: 10.1016/j.bbcan.2021.188665. Epub 2021 Dec 9. PMID 34896258
- [Background] Pinquart M, Duberstein PR. Depression and cancer mortality: a meta-analysis. Psychol Med. 2010 Nov;40(11):1797-810. doi: 10.1017/S0033291709992285. Epub 2010 Jan 20. PMID 20085667
- [Background] Macek P, Biskup M, Terek-Derszniak M, Stachura M, Krol H, Gozdz S, Zak M. Optimal Body Fat Percentage Cut-Off Values in Predicting the Obesity-Related Cardiovascular Risk Factors: A Cross-Sectional Cohort Study. Diabetes Metab Syndr Obes. 2020 May 12;13:1587-1597. doi: 10.2147/DMSO.S248444. eCollection 2020. PMID 32494175
- [Background] Battelino T, Danne T, Bergenstal RM, Amiel SA, Beck R, Biester T, Bosi E, Buckingham BA, Cefalu WT, Close KL, Cobelli C, Dassau E, DeVries JH, Donaghue KC, Dovc K, Doyle FJ 3rd, Garg S, Grunberger G, Heller S, Heinemann L, Hirsch IB, Hovorka R, Jia W, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Levine B, Mayorov A, Mathieu C, Murphy HR, Nimri R, Norgaard K, Parkin CG, Renard E, Rodbard D, Saboo B, Schatz D, Stoner K, Urakami T, Weinzimer SA, Phillip M. Clinical Targets for Continuous Glucose Monitoring Data Interpretation: Recommendations From the International Consensus on Time in Range. Diabetes Care. 2019 Aug;42(8):1593-1603. doi: 10.2337/dci19-0028. Epub 2019 Jun 8. PMID 31177185
- [Background] Advani A. Positioning time in range in diabetes management. Diabetologia. 2020 Feb;63(2):242-252. doi: 10.1007/s00125-019-05027-0. Epub 2019 Nov 7. PMID 31701199
- [Background] Liu Y, Pettersson E, Schandl A, Markar S, Johar A, Lagergren P. Dispositional optimism and all-cause mortality after esophageal cancer surgery: a nationwide population-based cohort study. Support Care Cancer. 2022 Nov;30(11):9461-9469. doi: 10.1007/s00520-022-07311-z. Epub 2022 Aug 11. PMID 35953730
- [Background] Thong MS, Kaptein AA, Vissers PA, Vreugdenhil G, van de Poll-Franse LV. Illness perceptions are associated with mortality among 1552 colorectal cancer survivors: a study from the population-based PROFILES registry. J Cancer Surviv. 2016 Oct;10(5):898-905. doi: 10.1007/s11764-016-0536-5. Epub 2016 Mar 19. PMID 26995005
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Mielnik M, Szudy-Szczyrek A, Homa-Mlak I, Mlak R, Podgajna-Mielnik M, Goracy A, Malecka-Massalska T, Hus M. The Clinical Relevance of Selected Cytokines in Newly Diagnosed Multiple Myeloma Patients. Biomedicines. 2023 Nov 9;11(11):3012. doi: 10.3390/biomedicines11113012. PMID 38002012
- [Background] Nachbaur DM, Herold M, Maneschg A, Huber H. Serum levels of interleukin-6 in multiple myeloma and other hematological disorders: correlation with disease activity and other prognostic parameters. Ann Hematol. 1991 Feb-Mar;62(2-3):54-8. doi: 10.1007/BF01714900. PMID 2031968
- [Background] Ludwig H, Nachbaur DM, Fritz E, Krainer M, Huber H. Interleukin-6 is a prognostic factor in multiple myeloma. Blood. 1991 Jun 15;77(12):2794-5. No abstract available. PMID 2043775
- [Background] Jasrotia S, Gupta R, Sharma A, Halder A, Kumar L. Cytokine profile in multiple myeloma. Cytokine. 2020 Dec;136:155271. doi: 10.1016/j.cyto.2020.155271. Epub 2020 Sep 8. PMID 32916474
- [Background] Esmaeilzadeh Z, Kheradmand F, Rasmi Y, Khadem-Ansari M. Serum levels of IL-6, TNF-α, and YKL-40 in patients with stage I multiple myeloma. J Res Appl Basic Med Sci Res Appl Basic Med Sci. 2020;6(3):160-166.
- [Background] Gu J, Huang X, Zhang Y, Bao C, Zhou Z, Jin J. Cytokine profiles in patients with newly diagnosed multiple myeloma: Survival is associated with IL-6 and IL-17A levels. Cytokine. 2021 Feb;138:155358. doi: 10.1016/j.cyto.2020.155358. Epub 2020 Nov 10. PMID 33183958
- [Background] Tsubaki M, Komai M, Itoh T, Imano M, Sakamoto K, Shimaoka H, Ogawa N, Mashimo K, Fujiwara D, Takeda T, Mukai J, Sakaguchi K, Satou T, Nishida S. Inhibition of the tumour necrosis factor-alpha autocrine loop enhances the sensitivity of multiple myeloma cells to anticancer drugs. Eur J Cancer. 2013 Nov;49(17):3708-17. doi: 10.1016/j.ejca.2013.07.010. Epub 2013 Aug 7. PMID 23932230
- [Background] Gervas J, Pocovi M, Giraldo P. Proinflammatory Cytokines Profile in Monoclonal Gammopathies Related to Pathogenesis of Bone Disease. Blood. 2009;114(22):4913-4913. doi:10.1182/blood.V114.22.4913.4913
- [Background] Jourdan M, Tarte K, Legouffe E, Brochier J, Rossi JF, Klein B. Tumor necrosis factor is a survival and proliferation factor for human myeloma cells. Eur Cytokine Netw. 1999 Mar;10(1):65-70. PMID 10210775
- [Background] Jurisic V, Colovic M. Correlation of sera TNF-alpha with percentage of bone marrow plasma cells, LDH, beta2-microglobulin, and clinical stage in multiple myeloma. Med Oncol. 2002;19(3):133-9. doi: 10.1385/MO:19:3:133. PMID 12482123
- [Background] Shapiro-Shelef M, Calame K. Plasma cell differentiation and multiple myeloma. Curr Opin Immunol. 2004 Apr;16(2):226-34. doi: 10.1016/j.coi.2004.02.001. PMID 15023417
- [Background] Tian T, Wang M, Ma D. TNF-alpha, a good or bad factor in hematological diseases? Stem Cell Investig. 2014 Jun 1;1:12. doi: 10.3978/j.issn.2306-9759.2014.04.02. eCollection 2014. PMID 27358858
- [Background] Spath F, Wibom C, Krop EJM, Santamaria AI, Johansson AS, Bergdahl IA, Hultdin J, Vermeulen R, Melin B. Immune marker changes and risk of multiple myeloma: a nested case-control study using repeated pre-diagnostic blood samples. Haematologica. 2019 Dec;104(12):2456-2464. doi: 10.3324/haematol.2019.216895. Epub 2019 Apr 4. PMID 30948485
- [Background] Ribas C, Colleoni GW, Felix RS, Regis Silva MR, Caballero OL, Brait M, Bordin JO. p16 gene methylation lacks correlation with angiogenesis and prognosis in multiple myeloma. Cancer Lett. 2005 May 26;222(2):247-54. doi: 10.1016/j.canlet.2004.09.038. Epub 2004 Nov 11. PMID 15863274
- [Background] Gkotzamanidou M, Christoulas D, Souliotis VL, Papatheodorou A, Dimopoulos MA, Terpos E. Angiogenic cytokines profile in smoldering multiple myeloma: no difference compared to MGUS but altered compared to symptomatic myeloma. Med Sci Monit. 2013 Dec 20;19:1188-94. doi: 10.12659/MSM.889752. PMID 24355943
- [Background] Palta A, Kaur M, Tahlan A, Dimri K. Evaluation of Angiogenesis in Multiple Myeloma by VEGF Immunoexpression and Microvessel Density. J Lab Physicians. 2020 Mar;12(1):38-43. doi: 10.1055/s-0040-1714933. Epub 2020 Jul 24. PMID 32792792
- [Background] Rapp K, Schroeder J, Klenk J, Ulmer H, Concin H, Diem G, Oberaigner W, Weiland SK. Fasting blood glucose and cancer risk in a cohort of more than 140,000 adults in Austria. Diabetologia. 2006 May;49(5):945-52. doi: 10.1007/s00125-006-0207-6. Epub 2006 Mar 24. PMID 16557372
- [Background] Tentolouris A, Ntanasis-Stathopoulos I, Eleftheriadou I, Malandrakis P, Tzeravini E, Gavriatopoulou M. Diabetes mellitus and multiple myeloma; common features of two distinct entities. Diabetes Metab Res Rev. 2022 Jul;38(5):e3535. doi: 10.1002/dmrr.3535. Epub 2022 May 25. PMID 35555946
- [Background] Thordardottir M, Lindqvist EK, Lund SH, Costello R, Burton D, Korde N, Mailankody S, Eiriksdottir G, Launer LJ, Gudnason V, Harris TB, Landgren O, Kristinsson SY. Obesity and risk of monoclonal gammopathy of undetermined significance and progression to multiple myeloma: a population-based study. Blood Adv. 2017 Nov 1;1(24):2186-2192. doi: 10.1182/bloodadvances.2017007609. eCollection 2017 Nov 14. PMID 29296866
- [Background] Liu L, Grandhi N, Wang M, et al. Association between excess body mass index trajectory and change in monoclonal protein level in patients diagnosed with monoclonal gammopathy of undetermined significance. J Clin Oncol. 2023;41(16_suppl):10538-10538. doi:10.1200/JCO.2023.41.16_suppl.10538
- [Background] Wallin A, Larsson SC. Body mass index and risk of multiple myeloma: a meta-analysis of prospective studies. Eur J Cancer. 2011 Jul;47(11):1606-15. doi: 10.1016/j.ejca.2011.01.020. Epub 2011 Feb 25. PMID 21354783
- [Background] Veld J, O'Donnell EK, Reagan MR, Yee AJ, Torriani M, Rosen CJ, Bredella MA. Abdominal adipose tissue in MGUS and multiple myeloma. Skeletal Radiol. 2016 Sep;45(9):1277-83. doi: 10.1007/s00256-016-2425-4. Epub 2016 Jun 25. PMID 27344672
- [Background] Teras LR, Kitahara CM, Birmann BM, Hartge PA, Wang SS, Robien K, Patel AV, Adami HO, Weiderpass E, Giles GG, Singh PN, Alavanja M, Beane Freeman LE, Bernstein L, Buring JE, Colditz GA, Fraser GE, Gapstur SM, Gaziano JM, Giovannucci E, Hofmann JN, Linet MS, Neta G, Park Y, Peters U, Rosenberg PS, Schairer C, Sesso HD, Stampfer MJ, Visvanathan K, White E, Wolk A, Zeleniuch-Jacquotte A, de Gonzalez AB, Purdue MP. Body size and multiple myeloma mortality: a pooled analysis of 20 prospective studies. Br J Haematol. 2014 Sep;166(5):667-76. doi: 10.1111/bjh.12935. Epub 2014 May 23. PMID 24861847
- [Background] Makris A, Pagkali A, Nikolousis E, Filippatos TD, Agouridis AP. High-density lipoprotein cholesterol and multiple myeloma: A systematic review and meta-analysis. Atheroscler Plus. 2023 Sep 21;54:7-13. doi: 10.1016/j.athplu.2023.09.003. eCollection 2023 Dec. PMID 37780686
- [Background] Tavori H, Ormseth MJ, Lilley JS, Papen CR, May-Zhang LS, Davies SS, Linton MF, Fazio S. Progressively decreasing plasma high-density lipoprotein cholesterol levels preceding diagnosis of smoldering myeloma. J Clin Lipidol. 2020 May-Jun;14(3):293-296. doi: 10.1016/j.jacl.2020.04.001. Epub 2020 Apr 13. PMID 32376310
- [Background] Liang L, Li J, Fu H, Liu X, Liu P. Identification of High Serum Apolipoprotein A1 as a Favorable Prognostic Indicator in Patients with Multiple Myeloma. J Cancer. 2019 Aug 27;10(20):4852-4859. doi: 10.7150/jca.31357. eCollection 2019. PMID 31598156
- [Background] Yazdani R, Marefati H, Shahesmaeili A, Nakhaei S, Bagheri A, Dastoorpoor M. Effect of Aerobic Exercises on Serum Levels of Apolipoprotein A1 and Apolipoprotein B, and Their Ratio in Patients with Chronic Obstructive Pulmonary Disease. Tanaffos. 2018 Feb;17(2):82-89. PMID 30627178
- [Background] Hofmann JN, Mailankody S, Korde N, Wang Y, Tageja N, Costello R, Zingone A, Hultcrantz M, Pollak MN, Purdue MP, Landgren O. Circulating Adiponectin Levels Differ Between Patients with Multiple Myeloma and its Precursor Disease. Obesity (Silver Spring). 2017 Aug;25(8):1317-1320. doi: 10.1002/oby.21894. Epub 2017 Jun 11. PMID 28602036
- [Background] Fowler JA, Lwin ST, Drake MT, Edwards JR, Kyle RA, Mundy GR, Edwards CM. Host-derived adiponectin is tumor-suppressive and a novel therapeutic target for multiple myeloma and the associated bone disease. Blood. 2011 Nov 24;118(22):5872-82. doi: 10.1182/blood-2011-01-330407. Epub 2011 Sep 8. PMID 21908434
- [Background] Dalamaga M, Christodoulatos GS. Adiponectin as a biomarker linking obesity and adiposopathy to hematologic malignancies. Horm Mol Biol Clin Investig. 2015 Jul;23(1):5-20. doi: 10.1515/hmbci-2015-0016. PMID 26057219
- [Background] Kriketos AD, Gan SK, Poynten AM, Furler SM, Chisholm DJ, Campbell LV. Exercise increases adiponectin levels and insulin sensitivity in humans. Diabetes Care. 2004 Feb;27(2):629-30. doi: 10.2337/diacare.27.2.629. No abstract available. PMID 14747265
- [Background] Vuong E, Nothling J, Lombard C, Jewkes R, Peer N, Abrahams N, Seedat S. Peripheral adiponectin levels in anxiety, mood, trauma- and stressor-related disorders: A systematic review and meta-analysis. J Affect Disord. 2020 Jan 1;260:372-409. doi: 10.1016/j.jad.2019.09.050. Epub 2019 Sep 11. PMID 31539673